CLINICAL TRIAL: NCT06954311
Title: Therapeutic Drug Monitoring for Biological Therapy in Pediatric Inflammatory Bowel Disease: a Prospective Non-interventional Multicentric Study
Brief Title: Therapeutic Drug Monitoring for Biological Therapy in Pediatric Inflammatory Bowel Disease
Acronym: TDMpIBD
Status: Recruiting | Type: Observational
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Other Study IDs: TDMpIBD (1126/2024)
Record Dates: First submitted 2025-04-07; First posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-03

CONDITIONS: Ulcerative Colitis (UC); IBD-unclassified (IBD-U)
Keywords: IBD; Pediatric; Biologicals; Infliximab; Adalimumab; Vedolizumab; Ustekinumab
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Infliximab Group: those who receive Infliximab
- Adalimumab Group: those who receive Adalimumab
- Vedolizumab Group: those who receive Vedolizumab
- Ustekinumab Group: those who receive Ustekinumab

SUMMARY:
Inflammatory Bowel Diseases (IBD), which include Crohn's disease (CD), ulcerative colitis (UC), and the unclassified form referred to as indeterminate colitis, are most commonly diagnosed during adolescence and early adulthood. In recent decades, an increasing incidence of IBD has been observed in this age group.

A wide range of immunomodulatory agents, from corticosteroids to monoclonal antibodies, are now available for the treatment of IBD. These antibodies, known as biologics, target, for example, tumor necrosis factor-alpha (TNF-α; e.g., infliximab and adalimumab), integrin α4β7 (vedolizumab), or interleukin-12/23 (ustekinumab). While infliximab and adalimumab are approved for pediatric use in CD and UC, vedolizumab is only approved for moderate-to-severe UC from the age of 16, and ustekinumab is not approved for pediatric use at all. Nevertheless, vedolizumab and ustekinumab are frequently used off-label in cases of treatment failure with approved therapies, as efficacy has been demonstrated in adult IBD patients, and since 2015, increasing pediatric literature has emerged on their use.

To facilitate appropriate dose adjustment in pediatric clinical practice, biologic therapies can be monitored through measurement of drug trough levels. Current pediatric guidelines already recommend incorporating therapeutic drug monitoring (TDM) of infliximab and adalimumab in the management of CD and UC. Studies on TDM for vedolizumab and ustekinumab have so far been conducted almost exclusively in adult IBD patients, where improved treatment responses have also been demonstrated.

The presented research is a prospective, non-interventional observational study involving pediatric IBD patients at multiple Austrian pediatric gastroenterology centers. The study duration is five years. The aim is to include at least 40 patients receiving induction and maintenance therapy with infliximab or adalimumab, and 20 patients treated with vedolizumab or ustekinumab during both treatment phases. The primary objective is to gain a better understanding of the pharmacokinetic dynamics of these biologics and the associated treatment response in pediatric settings. Data will be collected exclusively from routine clinical assessments. No additional study-related visits or interventions are planned.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients with an Inflammatory Bowel Disease (Crohn's disease, ulcerative colitis, and IBD-unclassified) being under 18 years of age
* Treatment with Infliximab, Adalimumab, Vedolizumab, or Ustekinumab during induction or maintenance phase

Exclusion Criteria:

-- Patients with primary (congenital) immunodeficiency

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients with IBD under 18 years of age (Crohn's disease, ulcerative colitis, and IBD-unclassified) with Treatment withInfliximab, Adalimumab, Vedolizumab, or Ustekinumab during induction or maintenance phase.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2030-02-17 (Estimated); Study Completion 2030-02-17 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic Evaluation of Plasma Level of Biological Therapy | Plasma Levels will be assessed at Baseline and approximately at Weeks 2, 6, 14, 22, 30, 38, 46, and 54 during routine follow-up visits. Actual timing may vary slightly due to the non-interventional nature of the study.
  Plasma levels of Infliximab, Adalimumab, Vedolizumab, and Ustekinumab will be assessed during routine follow-up visits, provided that such measurements are clinically indicated, in accordance with the non-interventional nature of the study design. The levels are measured in µg/ml.

SECONDARY OUTCOMES:
Time Course of Disease Activity (clinical assessments) | Clinical outcome scores will be assessed at Baseline and approximately at Weeks 2, 6, 14, 22, 30, 38, 46, and 54 during routine follow-up visits. Actual timing may vary slightly due to the non-interventional nature of the study
  Disease activity is assessed using validated clinical scoring systems. In patients with Crohn's disease, the weighted Pediatric Crohn's Disease Activity Index (wPCDAI) is applied, which ranges from 0 to 125 points; higher scores indicate increased disease activity. For patients with ulcerative colitis, the Pediatric Ulcerative Colitis Activity Index (PUCAI) is used, with a scoring range of 0 to 85 points-again, higher values reflect greater disease severity.
Time course of Disease Activity (laboratory assessments) | Calprotectin will be assessed at Baseline and approximately at Weeks 2, 6, 14, 22, 30, 38, 46, and 54 during routine follow-up visits. Actual timing may vary slightly due to the non-interventional nature of the study
  Disease activity is assessed by measuring fecal calprotectin levels, a biomarker indicative of intestinal inflammation. Elevated levels correlate with increased disease activity. Calprotectin is quantified in µg/g of stool, with values below 20.0 µg/g considered within the normal range. Measurements are performed using a standardized assay in the routine clinical laboratory.
Development of anti-drug antibodies during Biological Therapy | Anti-drug antibody Levels will be assessed at Baseline and approximately at Weeks 2, 6, 14, 22, 30, 38, 46, and 54 during routine follow-up visits. Actual timing may vary slightly due to the non-interventional nature of the study.
  Each time plasma levels of Infliximab, Adalimumab, Vedolizumab, or Ustekinumab are measured, the same laboratory also assesses the presence of anti-drug antibodies. If detectable, these antibodies will be quantified and reported in ng/mL. The presence of elevated anti-drug antibody levels has been linked to reduced treatment efficacy and an increased risk of therapeutic failure. The probability of developing anti-drug antibodies is relatively low; therefore, multiple time points are assessed to ensure accurate detection and monitoring over the course of treatment.

CONTACTS AND LOCATIONS:
Locations (10):
- Austria (10):
  - Landeskrankenhaus Feldkirch, Feldkirch
  - Universitätsklinikum Graz / Medizinische Universität Graz, Graz
  - Medical University of Innsbruck, Innsbruck
  - Klinikum Klagenfurt, Klagenfurt
  - Kepler Universitätsklinikum Linz, Linz
  - Paracelsus Medizinische Privatuniversität, Salzburg
  - St. Anna Kinderspital, Vienna
  - Universitätsklinik für Kinder- und Jugendheilkunde, Vienna
  - Klinik Donaustadt, Vienna
  - Landeskrankenhaus Villach, Villach

IPD SHARING:
Plan to Share IPD: Undecided